CLINICAL TRIAL: NCT03388190
Title: METIMMOX: Colorectal Cancer METastasis - Shaping Anti-tumor IMMunity by OXaliplatin
Acronym: METIMMOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: Trondheim University Hospital (Other); Haukeland University Hospital (Other); Hospital of Southern Norway Trust (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Prof Dr Anne Hansen Ree, Professor, MD PhD, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9M8; 2017-001845-29 (EudraCT Number)
Record Dates: First submitted 2017-12-08; First posted 2018-01-02 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal; Cancer; Neoplasm; Nivolumab; Fluorouracil; Metastatic; Oxaliplatin; Leucovorin
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Intervention Model Description: The METIMMOX study is a multicenter open-label randomized phase 2 trial in first-line treatment of MSS/pMMR-mCRC using the standard-of-care Nordic FLOX regimen (control arm) or sequential therapy with the Nordic FLOX regimen and nivolumab (experimental arm), to investigate whether the experimental arm shows superiority in PFS, safety, tolerability, and QoL.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): The control arm will consist of intermittent treatment with the Nordic FLOX regimen in terms of 8 cycles before break until disease progression, when therapy is reintroduced and administered for another 8 cycles before a new break. This schedule will be continued until progressive disease on ongoing therapy (PFS), intolerable toxicity, withdrawal of consent, or death, whichever occurs first.
  Interventions: Drug: FLOX
- Experimental Arm (Experimental): The experimental arm will consist of repeat 2 cycles of the Nordic FLOX regimen followed by 2 cycles of nivolumab for a total of 8 individual cycles before break until disease progression, when therapy is reintroduced and administered for another total of 8 individual cycles before a new break. This schedule will be continued until progressive disease on ongoing therapy (PFS), intolerable toxicity, withdrawal of consent, or death, whichever occurs first.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — FLOX: Intravenous oxaliplatin 85 mg/m2 on day 1; bolus 5-fluorouracil 500 mg/m2 and bolus Leucovorin on days 1 and 2; IV administration every 2 weeks.
  Nivolumab: 240 mg flat dose; IV administration every 2 weeks.
  Other Names: Oxaliplatin; 5-fluorouracil; Leucovorin
  Arms: Experimental Arm
Drug: FLOX — FLOX: Intravenous oxaliplatin 85 mg/m2 on day 1; bolus 5-fluorouracil 500 mg/m2 and bolus Leucovorin on days 1 and 2; IV administration every 2 weeks.
  Other Names: Oxaliplatin; 5-fluorouracil; Leucovorin
  Arms: Control Arm

SUMMARY:
This study aims to determine the efficacy, safety, and tolerability of the sequential addition of immune-modulating therapy to standard-of-care therapy of microsatellite-stable (MSS)/mismatch repair-proficient (pMMR) metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
Hypothesis: Patients with MSS/pMMR-mCRC harbor tumor that can be transformed into an immunogenic disease by short-course oxaliplatin-based therapy, and may thereby benefit from the addition of immune-modulating therapy to improve outcome of the current oxaliplatin-based standard-of-care.

Primary objective: To determine progression-free survival (PFS), in terms of failure of treatment strategy, of sequential treatment with the Nordic FLOX (5-Fluorouracil, oxaliplatin and leucovorin) regimen and nivolumab compared with the standard-of-care Nordic FLOX regimen in previously untreated MSS/pMMR-mCRC.

Secondary objectives: To determine safety and tolerability of sequential treatment with the Nordic FLOX regimen and nivolumab compared with the standard-of-care Nordic FLOX regimen. To monitor and compare quality-of-life (QoL) alterations during therapy courses.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically verified CRC adenocarcinoma (also comprising the mucinous adenocarcinoma and signet-ring cell carcinoma entities).
* Patient is ambulatory with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patient has radiologically measurable metastatic disease.
* Patient has an intra-abdominal metastatic lesion that can be biopsied.
* Patient has not had previous systemic therapy for the metastatic disease.
* Patient is eligible for the Nordic FLOX regimen.
* Patient has the following laboratory values, as measured in serum/plasma within 14 days prior to study entry, indicative of adequate organ function:

  * Hemoglobin at least 10.0 g/dL.
  * Neutrophils at least 1.5 x109/L (without current use of colony-stimulating factors).
  * Platelets at least 100 x109/L.
  * C-reactive protein (CRP) less than 60 mg/L.
  * Aspartate transaminase (AST)/Alanine transaminase (ALT) no higher than 2xULN when patient does not have metastatic disease in the liver or no higher than 5xULN when patient has metastatic disease in the liver.
  * Bilirubin no higher than 1.5x ULN when patient does not have metastatic disease in the liver or no higher than 2x upper limit of normal (ULN) when patient has metastatic disease in the liver.
  * Albumin no lower than 30 g/L.
  * International Normalised Ratio (INR) within normal level.
  * Creatinine no higher than 1.5x ULN.
* Woman of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
* WOCBP will use an adequate method to avoid pregnancy for a period of 26 weeks (which includes the required 30 days plus the time required for nivolumab to undergo five half-lives) after the last therapy dose, irrespective of study arm.
* Woman is not breastfeeding.
* Male who is sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a period of 26 weeks (which includes the required time to ensure duration of sperm turnover plus the time required for the investigational drugs to undergo five half-lives) after the last therapy dose, irrespective of study arm.
* Signed informed consent form (ICF) and expected cooperation of the patients for the treatment and follow-up must be obtained and documented according to International Conference on Harmonization (ICH) - Good Clinical Practice (GCP) and national/local regulations.

Exclusion Criteria:

* Patient has initially resectable metastatic disease for which neoadjuvant therapy is deemed superfluous.
* Patient does not consent to biopsy sampling.
* Patient has metastatic disease to lungs as the sole site.
* Patient has untreated or symptomatic brain metastasis (patient must be symptom-free without the use of corticosteroids).
* Patient experiences a period of less than 6 months since discontinuation of adjuvant oxaliplatin-containing chemotherapy.
* Patient is ineligible for full chemotherapy doses (100% doses) at start of study treatment.
* Patient has had radiation therapy against the only measurable lesion within 4 weeks of start of study treatment.
* Patient has any medical condition treated with anticoagulant medication that cannot be replaced by low molecular weight heparin during active study treatment.
* Patient has a nervous system disorder worse than Common Terminology Criteria for Adverse Events (CTCAE) grade 1.
* Patient has any medical condition that will preclude him/her from cancer immune-modulating therapy, such as:

  * Active or chronic hepatitis B or hepatitis C.
  * Known history of human immunodeficiency virus or acquired immunodeficiency-related illnesses.
  * Diagnosis of immunodeficiency or medical condition requiring systemic steroids or other forms of immunosuppressive therapy.
  * Autoimmune disease that has required systemic therapy within the past 2 years.
  * Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving study therapy.
  * Active infection or chronic infection requiring chronic suppressive antibiotics.
  * Known history of previous diagnosis of tuberculosis.
* Patient with current or prior use of immunosuppressive medication within 28 days before the first dose of study therapy, with the exceptions of intranasal corticosteroids or systemic corticosteroids at physiological doses that do not exceed 10mg/day of prednisone or an equivalent corticosteroid.
* Patient has any medical condition or needs to use medication, as listed in the Summary of Product characteristics (SmPC) of each Investigational Medical Product (IMP), that will preclude him/her from receiving treatment with IMP, such as:

  * Pernicious anemia or anemias due to vitamin B12 deficiency (SmPC-listed contraindications for folinic acid).
  * Other SmPC-listed contraindications for folinic acid and SmPC-listed contraindications for the other IMPs are covered by other exclusion criteria.
* Patient has undergone treatment with any IMP that may interfere with the study treatment within 4 weeks prior to first administration of study drug.
* Patient has known hypersensitivity to any of the study IMP components.
* Patient has ECOG performance status 2 or worse.
* Patient has serum/plasma CRP of 60 mg/L or higher.
* Patient does not meet the following requirements at baseline: adequate bone marrow function without current use of colony-stimulating factors (minimum values of neutrophils 1.5 x109/L, platelets 100 x109/L, hemoglobin 10 g/dL), adequate liver function (maximum values of AST/ALT 5x ULN and bilirubin 2x ULN; albumin value of 30 g/L or higher; INR within normal level), adequate renal function (maximum creatinine value of 1.5x ULN).
* Patient has history of other prior malignancy, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin, cervical cancer stage IB ( clinically visible lesion confined to cervix uteri), stage I prostate cancer considered not necessary to treat, and another malignancy that was treated with curative intent more than 5 years ago and has not relapsed later.
* Patient has significant cardiac, pulmonary, or other medical illness that would limit activity of daily life or survival.
* Patient is pregnant or breastfeeding.
* Patient has any other reason, in the opinion of Clinical Investigator, not to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary - progression-free survival (PFS) | Through study completion, an average of 15 months
  To determine PFS, in terms of failure of treatment strategy, on sequential treatment with the Nordic FLOX regimen and nivolumab compared with the standard-of-care Nordic FLOX regimen in previously untreated MSS mCRC.
  - PFS: radiologic assessment every 8 weeks (following 4 cycles of FLOX or the alternative 2 cycles each of FLOX and nivolumab), according to the Response Evaluation Criteria in Solid Tumors (RECIST) and the RECIST consensus guideline for assessment of response to immune-modulating therapies (iRECIST).

SECONDARY OUTCOMES:
Secondary 1 - Incidence (safety) and grading (tolerability) of treatment-related adverse events | Through study completion, an average of 15 months
  To determine the number of participants (incidence; safety) with treatment-related adverse events and their grading (tolerability), as assessed by CTCAE v4.0, of sequential treatment with the Nordic FLOX regimen and nivolumab compared with the standard-of-care Nordic FLOX regimen.
Secondary 2 - Objective response rate (ORR) | Through study completion, an average of 15 months
  To determine the percentage of patients with confirmed complete or partial response of sequential treatment with the Nordic FLOX regimen and nivolumab compared with the standard-of-care Nordic FLOX regimen.
Secondary 3 - Duration of response (DOR) | Through study completion, an average of 15 months
  To determine the time from the first documentation of a complete or partial response to disease progression of sequential treatment with the Nordic FLOX regimen and nivolumab compared with the standard-of-care Nordic FLOX regimen.
Secondary 4 - Secondary curative resection rate (SSCRR) | Through study completion, an average of 15 months
  To determine the percentage of patients with a confirmed resection of metastatic disease with microscopically free margin (R0) of sequential treatment with the Nordic FLOX regimen and nivolumab compared with the standard-of-care Nordic FLOX regimen.
Secondary 5 - Overall survival (OS) | Through study completion, an average of 15 months
  To determine the time from randomization to death of any cause of sequential treatment with the Nordic FLOX regimen and nivolumab compared with the standard-of-care Nordic FLOX regimen.
Secondary 6 - Quality-of-life (QoL) | Through study completion, an average of 15 months
  To monitor and compare QoL alterations during therapy courses using the consensus module EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life, 30 question version).
  Per the EORTC Scoring manual, the EORTC-QLQ-C30 uses 5 functional scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea and vomiting), a global health status/quality of life scale and a number of other questions which assess items such as dyspnoea, loss of appetite, insomnia, constipation and diarrhoea, as well as the perceived financial impact of having cancer. Scales range from 0 to 100, and a higher score means a higher response rate, where a high score on the functional or global health status questions represents a high or healthy level of functioning, quality of life or, alternatively, more symptoms or issues (symptom scale/items). [Scoring information summarised from the EORTC QLQ-C30 Scoring manual, 3rd edition]
Secondary 7 - Quality-of-life (QoL) | Through study completion, an average of 15 months
  To monitor and compare QoL alterations during therapy courses using the consensus module EORTC QLQ-CIPN20 (European Organisation for Research and Treatment of Cancer Quality of Life, 20 question Chemotherapy Induced Peripheral Neuropathy questionnaire).
  The EORTC QLQ-CIPN20 uses 20 questions assessing the quality of sensory, motor and autonomic symptoms on a 4-point Likert scale. Answers range from 1 (not at all) to 4 (very much). Patients indicate their perception of each item, and the scores are aggregated by quality, with a maximum of 32 points for motor, 36 for sensory, and either 12 (men) or 8 (women) in autonomic, where women would not answer a question about erectile function. Scores are then added together to give an overall score. The higher the score, the more symptoms the patient is experiencing.
Secondary 8 - Quality-of-life (QoL) | Through study completion, an average of 15 months
  To monitor and compare QoL alterations during therapy courses using the consensus module EQ-5D-5L (EuroQoL's 5-dimension, 5-level questionnaire).
  The EQ-5D-5L questionnaire is a "standardised measure of health status developed by the EuroQol group to provide a simple, generic measure of health for clinical and economic appraisal". The questionnaire uses 5 dimensions (5D) - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. There are 5 response levels: no issues, slight problems, moderate problems, severe problems and unable to function/extreme problems. These answers are geared appropriately to the specific questionbeing asked. Responses are coded from 0 for no problems to 5 for unable to function, and are combined to give a 5-digit code that will describe the patient's state of health. For example, 21111 would mean slight problems with mobility, but no other issues in the other dimensions. (summarised from the EQ-5D-5L user guide, v3.0).

OTHER OUTCOMES:
Tertiary - Cost estimate | Through study completion, an average of 15 months
  To compare costs for the resource use (in diagnostic work-up, treatment, and any adverse events) for the sequential therapy with that of the standard-of-care, applying a model specifically developed for CRC.
Exploratory 1 - Circulating biomarkers of cytotoxic T lymphocyte activity | Through study completion, an average of 15 months
  To monitor the individual patients' levels of PTEN (phosphatase and tensin homolog) phosphatase activity in peripheral blood mononuclear cells throughout study treatment.
Exploratory 2 - Circulating biomarkers of tumor response | Through study completion, an average of 15 months
  To monitor the individual patients' levels of plasma tumor DNA throughout study treatment.
Exploratory 3 - Circulating biomarkers of tumor immunogenic cell death (ICD) | Through study completion, an average of 15 months
  To monitor the individual patients' levels of serum/plasma immune proteins throughout study treatment.
Exploratory 4 - Functional MR (Magnetic Resonance) imaging biomarkers | Through study completion, an average of 15 months
  To monitor the individual patients' changes in liver/peritoneal functional MR signals throughout study treatment.
Exploratory 5 - Histologic and molecular tumor biomarkers | Through study completion, an average of 15 months
  To monitor the individual patients' changes in liver/peritoneal tissue composition throughout study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Ree, MD PhD, Principal Investigator — University Hospital, Akershus
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Hospital of Southern Norway, Department of Oncology, Kristiansand
  - Oslo University Hospital, Oslo
  - Akershus University Hospital, Oslo
  - St Olav's Hospital - Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No
No plan to share unrandomised, individual participant data with any researchers not involved in the study at the outset.

REFERENCES:
- [Background] Dueland S, Ree AH, Groholt KK, Saelen MG, Folkvord S, Hole KH, Seierstad T, Larsen SG, Giercksky KE, Wiig JN, Boye K, Flatmark K. Oxaliplatin-containing Preoperative Therapy in Locally Advanced Rectal Cancer: Local Response, Toxicity and Long-term Outcome. Clin Oncol (R Coll Radiol). 2016 Aug;28(8):532-9. doi: 10.1016/j.clon.2016.01.014. Epub 2016 Feb 14. PMID 26888115
- [Background] Flatmark K, Saelen MG, Hole KH, Abrahamsen TW, Fleten KG, Hektoen HH, Redalen KR, Seierstad T, Dueland S, Ree AH. Individual tumor volume responses to short-course oxaliplatin-containing induction chemotherapy in locally advanced rectal cancer - Targeting the tumor for radiation sensitivity? Radiother Oncol. 2016 Jun;119(3):505-11. doi: 10.1016/j.radonc.2016.02.020. Epub 2016 Mar 8. PMID 26968754
- [Background] Grovik E, Redalen KR, Storas TH, Negard A, Holmedal SH, Ree AH, Meltzer S, Bjornerud A, Gjesdal KI. Dynamic multi-echo DCE- and DSC-MRI in rectal cancer: Low primary tumor Ktrans and DeltaR2* peak are significantly associated with lymph node metastasis. J Magn Reson Imaging. 2017 Jul;46(1):194-206. doi: 10.1002/jmri.25566. Epub 2016 Dec 21. PMID 28001320
- [Background] Joranger P, Nesbakken A, Hoff G, Sorbye H, Oshaug A, Aas E. Modeling and validating the cost and clinical pathway of colorectal cancer. Med Decis Making. 2015 Feb;35(2):255-65. doi: 10.1177/0272989X14544749. Epub 2014 Jul 29. PMID 25073464
- [Background] Kalanxhi E, Hektoen HH, Meltzer S, Dueland S, Flatmark K, Ree AH. Circulating proteins in response to combined-modality therapy in rectal cancer identified by antibody array screening. BMC Cancer. 2016 Jul 26;16:536. doi: 10.1186/s12885-016-2601-x. PMID 27461255
- [Background] Meltzer S, Kalanxhi E, Hektoen HH, Dueland S, Flatmark K, Redalen KR, Ree AH. Systemic release of osteoprotegerin during oxaliplatin-containing induction chemotherapy and favorable systemic outcome of sequential radiotherapy in rectal cancer. Oncotarget. 2016 Jun 7;7(23):34907-17. doi: 10.18632/oncotarget.8995. PMID 27145458
- [Background] Ostrup O, Dagenborg VJ, Rodland EA, Skarpeteig V, Silwal-Pandit L, Grzyb K, Berstad AE, Fretland AA, Maelandsmo GM, Borresen-Dale AL, Ree AH, Edwin B, Nygaard V, Flatmark K. Molecular signatures reflecting microenvironmental metabolism and chemotherapy-induced immunogenic cell death in colorectal liver metastases. Oncotarget. 2017 Jul 18;8(44):76290-76304. doi: 10.18632/oncotarget.19350. eCollection 2017 Sep 29. PMID 29100312
- [Background] Ree AH, Flatmark K, Saelen MG, Folkvord S, Dueland S, Geisler J, Redalen KR. Tumor phosphatidylinositol 3-kinase signaling in therapy resistance and metastatic dissemination of rectal cancer: opportunities for signaling-adapted therapies. Crit Rev Oncol Hematol. 2015 Jul;95(1):114-24. doi: 10.1016/j.critrevonc.2015.01.003. Epub 2015 Jan 12. PMID 25624177
- [Background] Ree AH, Russnes HG, Heinrich D, Dueland S, Boye K, Nygaard V, Silwal-Pandit L, Ostrup O, Hovig E, Nygaard V, Rodland EA, Nakken S, Oien JT, Johansen C, Bergheim IR, Skarpeteig V, Sathermugathevan M, Sauer T, Lund-Iversen M, Beiske K, Nasser S, Julsrud L, Reisse CH, Ruud EA, Florenes VA, Hagene KT, Aas E, Luras H, Johnsen-Soriano S, Geitvik GA, Lingjaerde OC, Borresen-Dale AL, Maelandsmo GM, Flatmark K. Implementing precision cancer medicine in the public health services of Norway: the diagnostic infrastructure and a cost estimate. ESMO Open. 2017 May 2;2(2):e000158. doi: 10.1136/esmoopen-2017-000158. eCollection 2017. PMID 28761742
- [Background] Spindler KG, Boysen AK, Pallisgard N, Johansen JS, Tabernero J, Sorensen MM, Jensen BV, Hansen TF, Sefrioui D, Andersen RF, Brandslund I, Jakobsen A. Cell-Free DNA in Metastatic Colorectal Cancer: A Systematic Review and Meta-Analysis. Oncologist. 2017 Sep;22(9):1049-1055. doi: 10.1634/theoncologist.2016-0178. Epub 2017 Aug 4. PMID 28778958
- [Background] Tveit KM, Guren T, Glimelius B, Pfeiffer P, Sorbye H, Pyrhonen S, Sigurdsson F, Kure E, Ikdahl T, Skovlund E, Fokstuen T, Hansen F, Hofsli E, Birkemeyer E, Johnsson A, Starkhammar H, Yilmaz MK, Keldsen N, Erdal AB, Dajani O, Dahl O, Christoffersen T. Phase III trial of cetuximab with continuous or intermittent fluorouracil, leucovorin, and oxaliplatin (Nordic FLOX) versus FLOX alone in first-line treatment of metastatic colorectal cancer: the NORDIC-VII study. J Clin Oncol. 2012 May 20;30(15):1755-62. doi: 10.1200/JCO.2011.38.0915. Epub 2012 Apr 2. PMID 22473155
- [Derived] Ree AH, Saltyte Benth J, Hamre HM, Kersten C, Hofsli E, Guren MG, Sorbye H, Johansen C, Negard A, Bjornetro T, Nilsen HL, Berg JP, Flatmark K, Meltzer S. First-line oxaliplatin-based chemotherapy and nivolumab for metastatic microsatellite-stable colorectal cancer-the randomised METIMMOX trial. Br J Cancer. 2024 Jun;130(12):1921-1928. doi: 10.1038/s41416-024-02696-6. Epub 2024 Apr 25. PMID 38664577
- [Derived] Meltzer S, Negard A, Bakke KM, Hamre HM, Kersten C, Hofsli E, Guren MG, Sorbye H, Flatmark K, Ree AH. Early radiologic signal of responsiveness to immune checkpoint blockade in microsatellite-stable/mismatch repair-proficient metastatic colorectal cancer. Br J Cancer. 2022 Dec;127(12):2227-2233. doi: 10.1038/s41416-022-02004-0. Epub 2022 Oct 13. PMID 36229579